CLINICAL TRIAL: NCT03733223
Title: Relationships Among FVIII, t-PA/PAI-1, and MMP-9 Levels and Intracranial Hemorrhage Complications After Thrombolysis With Alteplase in Patients With Acute Ischemic Stroke: Protocol for a Multicenter Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); First Affiliated Hospital of Jinan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-YXB-002
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Stroke
Keywords: t-PA/PAI-1; MMP-9; FVIII; Alteplase; intracranial haemorrhage; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: The patients who were treated with Ateptidase had intracranial haemorrhage adverse reactions
  Interventions: Drug: Ateptidase
- control group: The patients who were treated with Ateptidase did not have intracranial haemorrhage adverse reactions.
  Interventions: Drug: Ateptidase

INTERVENTIONS:
Drug: Ateptidase — Treatment of ischemic stroke with Ateptidase

SUMMARY:
The primary aim of the study is to investigate the relationships among FVIII, t-PA/PAI-1, MMP-9 levels, and intracranial hemorrhage after thrombolysis with alteplase using a combined analysis.

DETAILED DESCRIPTION:
Patients with acute ischemic stroke treated with alteplase within 4.5 hours after the onset of stroke symptoms will be recruited in this study. All participants will be divided into two groups according to whether intracranial hemorrhage occurred within 3 days after treatment with alteplase for analysis. Differences in FVIII, t-PA/PAI-1, and MMP-9 levels before and after thrombolytic therapy will be examined in both groups. This study will be conducted at Zhujiang Hospital of Southern Medical University, Nanfang Hospital of Southern Medical University, and the First Affiliated Hospital of Jinan University.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke and within the time window of thrombolysis (Onset of symptoms no more than 4.5 hours )
* 18 y age 85 y•
* Symptoms of neurological deficits caused by cerebral infarction
* Informed consent form to confirm thrombolytic therapy have signed by patients or their family.

Exclusion Criteria:

* A history of major head trauma or stroke in the past 3 months
* Suspicious subarachnoid hemorrhage
* Arterial puncture at noncompressible site in the last week
* History of intracranial hemorrhage
* Intracranial neoplasm, arteriovenous malformation, or aneurysm
* Recent intracranial or intraspinal surgery
* Elevated blood pressure (systolic >185 mm Hg or diastolic >110 mm Hg)
* Active internal bleeding or Acute bleeding diathesis
* Platelet count <100×109·L-1
* Heparin received within 48 h resulting in aPTT above the upper limit of normal
* Current use of anticoagulant with INR >1.7 or PT >15 s
* Current use of thrombin inhibitors or factor Xa inhibitors
* Abnormal laboratory tests (eg, aPTT, INR, platelet count, ECT, TT, or appropriate factor Xa activity assays)
* Blood glucose concentration > 2.7 mmol/L
* CT demonstrates multilobar infarction (hypodensity >1/3 cerebral hemisphere)
* Mild cerebral infarction or rapid improvement of symptoms of cerebral infarction
* Symptoms of neurological impairment after seizures
* Major surgery or severe trauma in the past 2 weeks
* Gastrointestinal or urinary bleeding in the past 3 weeks
* History of myocardial infarction in the past 3 months
* Combine diseases that may affect outcomes,such as Anemia, hemophilia
* History of autoimmune disease or organ transplantation
* Pregnancy or breastfeeding women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke treated with Alteplase
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-10-12 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Intracranial hemorrhage | 3 days
  The occurrence of intracranial haemorrhage adverse reactions in ischemic stroke patients receiving thrombolytic therapy by alteplase

CONTACTS AND LOCATIONS:
Overall Officials: Shuai He, Doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang Y, Liao X, Zhao X, Wang DZ, Wang C, Nguyen-Huynh MN, Zhou Y, Liu L, Wang X, Liu G, Li H, Wang Y; China National Stroke Registry Investigators. Using recombinant tissue plasminogen activator to treat acute ischemic stroke in China: analysis of the results from the Chinese National Stroke Registry (CNSR). Stroke. 2011 Jun;42(6):1658-64. doi: 10.1161/STROKEAHA.110.604249. Epub 2011 Apr 21. PMID 21512182